CLINICAL TRIAL: NCT01047449
Title: Surgical and Pharmacological Novel Interventions to Improve Overall Results of Saphenous Vein Graft Patency in Coronary Artery Bypass Grafting Surgery: An International Multi-Center Randomized Controlled Clinical Trial
Brief Title: Improving the Results of Heart Bypass Surgery Using New Approaches to Surgery and Medication
Acronym: SUPERIORSVG
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Sunnybrook Health Sciences Centre (Other)
Collaborators: Hamilton Health Sciences Corporation (Other)
Responsible Party: Principal Investigator, Stephen E. Fremes, Head, Division of Cardiac & Vascular Surgery, Sunnybrook Health Sciences Centre
Allocation: Randomized | Model: Factorial | Masking: Quadruple | Purpose: Treatment
Other Study IDs: CANNeCTIN09-11
Record Dates: First submitted 2010-01-12; First posted 2010-01-13 (Estimated); Last update posted 2017-10-05 (Actual); Status verified 2017-10

CONDITIONS: Coronary Artery Disease
Keywords: saphenous vein graft patency; fish oil supplementation; coronary artery bypass surgery; coronary artery disease
MeSH Terms: conditions — Coronary Artery Disease

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes

ARMS (4):
- SVG harvest - conventional, placebo (Active Comparator)
  Interventions: Procedure: No-touch SVG harvest vs conventional SVG harvest technique; Dietary Supplement: Fish oil supplementation vs placebo
- SVG harvest - no-touch, fish oils (Experimental)
  Interventions: Procedure: No-touch SVG harvest vs conventional SVG harvest technique; Dietary Supplement: Fish oil supplementation vs placebo
- SVG harvest - no-touch, placebo (Placebo Comparator)
  Interventions: Procedure: No-touch SVG harvest vs conventional SVG harvest technique; Dietary Supplement: Fish oil supplementation vs placebo
- SVG harvest - conventional, fish oils (Active Comparator)
  Interventions: Procedure: No-touch SVG harvest vs conventional SVG harvest technique; Dietary Supplement: Fish oil supplementation vs placebo

INTERVENTIONS:
Procedure: No-touch SVG harvest vs conventional SVG harvest technique — Saphenous vein harvested using the pedicled (no-touch) technique or using the conventional technique. Fish oil supplements/placebo (1g taken orally twice daily for 1 year post-op)
Dietary Supplement: Fish oil supplementation vs placebo — Fish oil supplementation [1g tablets (55% fish oils - EPA:DHA 33%:22%)] taken twice daily for 1 year post-op
  Other Names: Ocean Nutrition Omega Pure fish oil capsules

SUMMARY:
Surgery for blocked arteries in the heart (coronary artery bypass grafting) can be accomplished using veins from the leg sewn onto the heart to provide an alternate path for blood flow, i.e. 'bypassing' the blockages. These veins themselves can block over time. This may result in part simply from the trauma from the surgery, in other words, by removing the vein from the leg and then sewing it to the heart. Another mechanism may be the abnormal metabolic processes within the body responsible for the plaque build-up of the heart arteries in the first place - this may lead to the blockages of the veins used for bypass. In the present era of heart bypass surgery, this incidence of veins blocking remains high despite advances in blood thinners and cholesterol medications. This study is designed to determine whether two new interventions may potentially reduce the incidence of blockages in the veins used for heart bypass surgery. One is a surgical technique significantly reducing the trauma associated with removing the leg vein prior to use as a bypass graft onto the heart. The second intervention is the use of a nutritional supplement before and after surgery which is composed of fish oils. The study will recruit sufficient patients to provide strong and relevant conclusions regarding both study questions. It will be highly applicable also because it will include approximately 1,550 patients from approximately 50 hospitals across many countries. We believe these techniques will result in significantly less vein blockages in patients one year after heart bypass surgery.

DETAILED DESCRIPTION:
Background: Saphenous vein grafts (SVG) remain the most widely used conduit for CABG. However, contemporary patency rates at one-year post CABG remain poor, despite optimal medical therapy. Recent trials (PREVENT IV) demonstrate that up to 45% of all patients have one or more SVG occluded at angiography one year post-CABG; up to 25% of all SVG are occluded at one year post-CABG angiography. Furthermore, patients with at least one SVG occluded had twice the incidence of perioperative MI, and thirteen times the composite endpoint of death, late MI or repeat revascularization at 12-18 months.

The proposed SUPERIOR SVG Trial is a prospective, international, multi-centre randomized controlled clinical trial (RCT). It utilizes a factorial design to elucidate the benefits of two interventions, one surgical and the other pharmacological, to improve saphenous vein graft patency after coronary artery bypass grafting surgery (CABG):

Surgical Arm: Does a novel atraumatic ("no touch") technique of pedicled saphenous vein graft (SVG) harvesting result in improved angiographic patency and clinical outcomes at 1 year, compared to conventional SVG harvesting techniques, in patients undergoing CABG.

Rationale: A Swedish cardiac surgical centre has published numerous studies demonstrating that harvesting the SVG with a cushion of surrounding fat and without vein graft distension, "no touch" technique, improved surrogate markers of vein preservation in operative specimens. Graft patency was superior in a single small RCT (8.5 year patency: "no touch" 90% vs. conventional 76%, p=0.01, adjusted OR 3.7, 95% CI 1.4-9.6, p=0.007).

Pharmacological Arm: Does N-3 polyunsaturated fatty acid (fish oil) oral supplementation result in improved angiographic patency and clinical outcomes at 1 year, compared to placebo, in patients undergoing CABG.

Rationale: In vivo studies showed levels of N-3 polyunsaturated fatty acids (PUFA; fish-oils) inversely correlate with the risk of coronary disease. Several large RCTs (more than 40,000 patients in aggregate) performed in diverse cardiovascular populations, have demonstrated moderate mortality benefits. A single RCT from the 90's found that that SVG patency was enhanced with fish oils.

Methods: Each patient will be randomized to a SVG harvested in the conventional fashion (open or endoscopic) or using the "no touch" technique (single-blinded). The pharmacological arm of the factorial design will have patients also randomized to fish-oil or placebo (double-blinded) starting prior to surgery and continuing for 1 year. The primary outcomes (Surgical Arm: proportion of study SVG grafts occluded; Pharmacological Arm: proportion of patients with ≥1 graft occluded) at 1 year CT angiography (window 9-15 months) will be compared between the treatment and control groups. Secondary endpoints include incidence of 50-99% study SVG stenosis at 1 year, adverse events and perioperative and 1 year clinical events (mortality, non-fatal MI, repeat revascularization).

A sample size of 615 patients/arm will provide adequate statistical power (Surgical Arm, Primary Outcome: study SVG graft occlusion, control event rate = 20%, no-touch event rate = 14%, RRR = 0.30, β = 0.2; Pharmacological Arm, Primary Outcome: patients with at least 1 graft occlusion, control event rate = 30%, fish oils event rate 22.5%, RRR = 0.25, β= 0.15). The total sample size has been increased 25% to 1550 patients as approximately 20% of recruited patients in angiographic trials fail to undergo follow-up angiography. Study patients will be enrolled over 39 months at 50 centers. Pilot funding has been secured from CIHR-CANNeCTIN to assess feasibility in 50 patients from 15 sites. A single interim analysis will be performed following completion of 50% of the CT angiograms, p<0.001.

ELIGIBILITY:
Inclusion Criteria:

1. Age > 18 years
2. Able to provide informed consent
3. Isolated CABG, non-emergent, on- or off-pump (cardiopulmonary bypass)
4. Primary or re-do CABG (if re-do, all previous grafts must be occluded)
5. Left ventricular ejection fraction >20%
6. Require at least one SVG as part of revascularization strategy
7. Creatinine clearance of at least 30ml/min or higher

Exclusion Criteria:

1. Unable to use greater SV due to previous vein stripping or poor quality on mandatory preoperative Duplex study and vein mapping
2. Contraindication to receiving follow-up 64-slice cardiac CT angiography (allergy to contrast dye, renal failure with a creatinine >180 µmol/L, uncontrolled atrial fibrillation precluding proper gating of study)
3. Pregnant women, or women of child-bearing age
4. Allergy to fish oil/fish products, and non-medicinal ingredients of the study product (corn oil,soybean oil,gelatin,glycerol, or carob colouring)
5. Already taking fish oil supplements regularly (daily use in past 30 days)
6. Congenital or acquired coagulation disorders
7. Patients considered to be of excessive risk of wound infection according to the clinical judgement of the site surgical investigator.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 250 (Actual)
Dates: Start 2011-07; Primary Completion 2015-08 (Actual); Study Completion 2017-03-21 (Actual)

PRIMARY OUTCOMES:
Surgical Arm: Proportion of study SVGs which are totally occluded on cardiac CT angiography at 1-year post-CABG and death due to CV or unknown causes. | 1 year post-operative
Pharmacological Arm: Proportion of patients with ≥1 graft (saphenous or arterial) totally (100%) occluded on cardiac CT angiography at 1-year post-CABG and death due to CV or unknown causes, comparing the fish-oil to placebo groups. | 1-year post-operative

SECONDARY OUTCOMES:
Surgical Arm: i. To determine whether the "no touch" technique of SVG harvesting results in a lower proportion of study SVGs that have a significant stenosis (50-99%) on 1-year post-CABG angiography compared to conventional SVG harvesting techniques. | 1 year post-operavtive
Surgical Arm: ii. To determine whether the incidence and severity of adverse SVG harvesting events at 1-yr post-CABG (infection, haematoma, swelling, neuropathy, quality of life measures) are similar between the "no touch" and conventional groups. | 1-year post-operative
Surgical Arm: iii. The incidence of the composite of non-fatal MI (new definition), all-cause mortality, and repeat revascularization (redo CABG or PCI) perioperatively ( major adverse cardiac events ,MACE ) and stroke at 1 yr is lowe | 1-year post-operative
Pharmacological Arm: i. To determine whether fish oil supplementation results in a lower proportion of patients with ≥1 graft with a significant (50-99%) stenosis at 1-year post-CABG angiography, compared to those who received placebo. | 1-year post-operative
Pharmacological Arm: ii. The incidence of the composite of n-fatal MI (new definition), all-cause mortality, and repeat revascularization (redo CABG or PCI) perioperatively ( major adverse cardiac events ,MACE ) and stroke at 1 yr i | 1-year post-operative

CONTACTS AND LOCATIONS:
Overall Officials: Stephen Fremes, MD, Principal Investigator — Sunnybrook Health Sciences Centre
Locations (1):
- Sunnybrook Health Sciences Centre, Toronto, Ontario, Canada

REFERENCES:
- [Derived] Deb S, Singh SK, de Souza D, Chu MWA, Whitlock R, Meyer SR, Verma S, Jeppsson A, Al-Saleh A, Brady K, Rao-Melacini P, Belley-Cote EP, Tam DY, Devereaux PJ, Novick RJ, Fremes SE; SUPERIOR SVG Study Investigators. SUPERIOR SVG: no touch saphenous harvesting to improve patency following coronary bypass grafting (a multi-Centre randomized control trial, NCT01047449). J Cardiothorac Surg. 2019 May 2;14(1):85. doi: 10.1186/s13019-019-0887-x. PMID 31046806